CLINICAL TRIAL: NCT05007899
Title: Alternate Day Versus Daily Oral Iron Therapy in Adolescents With Iron Deficiency Anemia and Heavy Menstrual Bleeding: A Feasibility Trial
Brief Title: Alternate Day Versus Daily Oral Iron Therapy in Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jacquelyn Powers, MD, MS, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H - 46363
Record Dates: First submitted 2021-07-20; First posted 2021-08-17 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Iron Deficiency Anemia; Heavy Menstrual Bleeding; Abnormal Uterine Bleeding
MeSH Terms: conditions — Anemia, Iron-Deficiency; Menorrhagia; Metrorrhagia | interventions — ferrous sulfate; Iron; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daily (Active Comparator): Patients receive standard regimen of ferrous sulfate 325 mg (65 mg elemental iron) once every morning.
  Interventions: Drug: Ferrous sulfate
- Alternate Day (Experimental): Patients receive ferrous sulfate 325 mg (65 mg elemental iron) once every other morning.
  Interventions: Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Ferrous sulfate — Alternate day dosing of ferrous sulfate
  Other Names: Fer-In-Sol; Feratab; Iron; Feosol

SUMMARY:
Iron deficiency anemia affects over half of girls and young women with heavy periods and is the most common cause of anemia worldwide. Most girls with heavy periods who also have iron deficiency anemia are prescribed iron to take by mouth every day by their doctor. There are some studies showing that taking iron every other day may actually help the iron be absorbed into the bloodstream better. This study is trying to compare how taking iron every other day compares to taking iron daily for treatment of anemia.

The goal of this clinical research study is to learn which of the two methods of care will be the best way for girls and young women with iron deficiency anemia to take iron supplementation.

DETAILED DESCRIPTION:
The research will be conducted at the following location(s):

Baylor College of Medicine, TCH: Texas Children's Hospital, and TCH: Texas Children's Hospital Clinic.

If patient appears to qualify for the study they will sign and date this consent form, and the doctor will confirm that they are eligible for the study. The patient will complete the following procedures:

* Medical history including prior hospitalizations, lab results, medications, diet, social and family history
* Physical Examination
* Blood samples: The patient will not have any extra blood draws (pokes) for this study. However, we will ask to take about 1/2 (0.5) teaspoons (3 mL) of extra blood for an extra research test when you have follow up blood test(s) in one month.

Patient will be on the study for 24 weeks (6 months),and will receive an information sheet about how to take iron to help it absorb in the stomach and on iron-rich foods.

There are 2 different treatments in this study. If a patient enrolls, they cannot choose which treatment to receive. Instead, they will be randomly assigned to one of the two treatments. That means there is a fifty percent chance they will receive iron medicine to take every day and a fifty percent chance they will receive iron medicine to take every other day.

ELIGIBILITY:
Inclusion Criteria:

1. Age 9 years or greater and less than age 22 years
2. Heavy menstrual bleeding, defined as a Pictorial Blood Assessment Chart (PBAC) Score >100
3. Iron deficiency anemia, defined as both hemoglobin <12 g/dL and ferritin <15 ng/mL within 7 days of enrollment.

Exclusion Criteria:

1. non-uterine cause of vaginal bleeding
2. pregnancy
3. chronic kidney disease
4. serology confirmed celiac disease
5. active gastrointestinal blood loss
6. active malignancy
7. inability to follow-up at Texas Children's Hospital
8. receipt of intravenous iron within 30 days prior to enrollment
9. allergy or known inability to tolerate oral iron

Ages: 9 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Must be born a female.
Enrollment: 13 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Powers, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Pavilion for Women, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily | Alternate Day
Started | 7 | 6
Completed | 5 | 2
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily | Alternate Day | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 13 [12 to 14] | 16 [14 to 18] | 14 [12 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
PBAC Score [Median (Inter-Quartile Range); unit: Scores of a scale] — PBAC = Pictorial Blood Assessment Chart. The PBAC is a pictorial tool used to assess menstrual blood loss. The minimum score is 0. There is no maximum score. Higher scores are worse. A total score is reported with no subscales. An "abnormal" PBAC, which is consistent with a diagnosis of heavy menstrual bleeding is a score greater or equal to 100.
  Scores of a scale | 455 [228 to 618] | 144 [120 to 700] | 325 [121 to 780]
Hemoglobin (g/dL) [Median (Inter-Quartile Range); unit: g/dL] | 6.8 [6.0 to 9.7] | 5.7 [5.0 to 9.8] | 6.3 [5.6 to 11.1]
Post transfusions hemoglobin (g/dL) [Median (Inter-Quartile Range); unit: g/dL] | 8.4 [7.7 to 10.95] | 7.7 [7.45 to 1028] | 8.2 [7.7 to 11.1]
Mean Corpuscular volume (MCV, fL) [Median (Inter-Quartile Range); unit: fl] | 80.8 [71.2 to 82.2] | 74.9 [67.3 to 83.3] | 78.5 [70.5 to 83.4]
Serum ferritin (ng/mL) [Median (Inter-Quartile Range); unit: ng/mL] | 4 [3 to 7] | 9.5 [4.5 to 10.75] | 5 [3 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Patients Enrolled.
Description: Percentage of eligible patients who consent to be enrolled in the study. A secure screening and enrollment log will be kept. Each screened patient will be categorized as either: ineligible, eligible but not approached, eligible and enrolled, eligible and declined. If the latter (eligible and declined), the reason for declining will also be obtained and noted in the study log.
Time Frame: At enrollment
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Patients: Primary outcome was the percentage of eligible patients approached for the study who consented to enroll.
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 20
Participants | 13

2. Secondary Outcome: Percentage of Enrolled Patients Who Agree to Continue in the Study After Randomization
Description: Percentage of patients who continue in study as compared to total number of enrolled patients. Information will be obtained from the study log.
Time Frame: At enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Daily | Alternate Day
Number analyzed (Participants) | 7 | 6
Participants | 7 | 6

3. Secondary Outcome: Retention as Measured by Visit Follow-up Adherence
Description: Percentage of enrolled patients that completed 12 weeks of the study.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Daily | Alternate Day
Number analyzed (Participants) | 7 | 6
Participants | 5 | 2

4. Secondary Outcome: Adherence
Description: Pill counts were performed as an objective measure of adherence. Subjects were given a specific number of pills for the duration of the study. At the 12 week visit they were asked to return any remaining pills, which were then counted and compared to the number of expected pills should be remaining, assuming 100% adherence. These numbers were used to calculate an estimate of adherence.
Time Frame: 12 week study visit
Measure: Median (Full Range); unit: % of pills consumed
Arm/Group | Daily | Alternate Day
Number analyzed (Participants) | 7 | 6
% of pills consumed | 65 [31 to 100] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Twelve weeks
Description: All-Cause Mortality, Serious Adverse Events, and Other (Gastrointestinal) Adverse Events were collected at the 12 week visit.
Arm/Group | Daily | Alternate Day
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 3/5 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily (N=5) | Alternate Day (N=2)
Heartburn (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT05007899/Prot_SAP_001.pdf